CLINICAL TRIAL: NCT01336803
Title: Pilot Differentiation of Bone Sarcomas and Osteomyelitis With Ferumoxytol-Enhanced MRI
Brief Title: Differentiation of Bone Sarcomas and Osteomyelitis With Ferumoxytol-Enhanced MRI
Acronym: Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heike E Daldrup-Link (Other)
Responsible Party: Sponsor-Investigator, Heike E Daldrup-Link, Professor of Radiology (General Radiology), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-20253(osteosarcoma); SU-04062011-7666 (Other: Stanford University); PEDSBONE0006 (Other: OnCore Number)
Record Dates: First submitted 2011-04-12; First posted 2011-04-18 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Bone Cancer; Chondrosarcoma; Ewing's Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Bone Necrosis; Bone Sarcoma; Osteomyelitis
MeSH Terms: conditions — Bone Neoplasms; Chondrosarcoma; Sarcoma, Ewing; Osteosarcoma; Rhabdomyosarcoma; Osteonecrosis; Osteomyelitis | interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feraheme (Experimental): Intravenous injection of Feraheme, 5 mg Fe/kg
  Interventions: Drug: Feraheme; Procedure: Magnetic Resonance Imaging (MRI) scan

INTERVENTIONS:
Drug: Feraheme — 5 mg/kg by intravenous (IV) administration
  Other Names: ferumoxytol
Procedure: Magnetic Resonance Imaging (MRI) scan — Standard of Care magnetic resonance imaging (MRI) scans using GE 1.5T and 3T MRI scanners/
  Other Names: Magnetic Resonance (MR) scan

SUMMARY:
This pilot trial studies the differentiation of bone sarcomas and osteomyelitis with ferumoxytol-enhanced magnetic resonance imaging (MRI). Imaging procedures that allow doctors to more accurately differentiate between malignant bone sarcomas and osteomyelitis may help in diagnosing patients correctly and may result in more timely treatment.

DETAILED DESCRIPTION:
BACKGROUND; In this study, T1, T2, and T2* represent parameters of magnetic resonance imaging (MRI).

The T1 relaxation time, also known as the spin-lattice relaxation time, is a measure of how quickly the net magnetization vector (NMV) recovers to its ground state in the direction of B0. T1 is assessed immediately post-contrast. A T1-weighted image (T1WI ) is one of the basic pulse sequences in MRI and demonstrates differences in the T1 relaxation times of tissues. A T1WI relies upon the longitudinal relaxation of a tissue's net magnetization vector (NMV).

T2 is a time constant for the decay of transverse magnetization arising from natural interactions at the atomic or molecular levels, and be considered the "natural" or "true" T2 of the tissue. However, in any nuclear magnetic resonance (NMR) experiment, transverse magnetization decays much faster than would be predicted by natural atomic and molecular mechanisms. Accordingly, T2 * is the time constant for the decay of transverse magnetization as observed in a tissue during a MRI scan, and be considered the"effective T2" (represented as T2*). T2* is always ≤ T2. In this study, T2 * is assessed after 24 hours.

OUTLINE:

Patients receive ferumoxytol intravenously (IV) and then undergo ferumoxytol-enhanced MRI up to 1 hour after infusion and up to 24 hours post-infusion.

PRIMARY OBJECTIVES:

* Establish magnetic resonance (MR) imaging characteristics of bone sarcomas and osteomyelitis based on their ferumoxytol-enhancement on relatively early post-contrast T1-weighted images.
* Establish MR imaging characteristics of bone sarcomas and osteomyelitis based on their ferumoxytol-enhancement on delayed postcontrast T2-weighted images.
* Establish T2-weighted MR imaging characteristics of iron-labeled mesenchymal stem cell (MSC) in osteonecrotic bone over time, before and after surgical core decompression and bone marrow implantation.
* Adding a second branch for patients who can not receive ferumoxytol but still getting the MRI exam. These patients will server as controls.

ELIGIBILITY:
INCLUSION CRITERIA

* Age 10 to 21 years
* Suspected or confirmed diagnosis of a bone sarcoma or osteomyelitis
* Informed consent with assent as appropriate.

EXCLUSION CRITERIA

* Contraindication to MRI
* Presence of metal implants
* Need for sedation or anesthesia
* Claustrophobia
* Hemosiderosis or hemochromatosis
* History of allergic reactions to similar compounds will be obtained and patients with positive history of allergic reactions will be excluded from the study
* Females who are pregnancy or nursing

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2023-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heike E Daldrup-Link, MD, Principal Investigator — Stanford University; Neyssa Marina, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Feraheme: Intravenous injection of Feraheme, 5 mg Fe/kg
  Feraheme: 5 mg Fe/kg by intravenous adminstration
  MR Scan: Standard of Care
Period: Overall Study
Arm/Group | Feraheme
Started | 21
Bone Sarcoma | 10
Osteomyelitis | 4
Lymphoma | 7
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Feraheme
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: T2* Relaxation Time of Bone Sarcomas and Osteomyelitis Subjects
Description: Differentiation of bone sarcomas and osteomyelitis with ferumoxytol-enhanced magnetic resonance imaging (MRI) was assessed as the difference of mean T2 * relaxation time of bone sarcoma and osteomyelitis subjects. The outcome is reported as the difference of the mean T2 * values, with standard deviation.
Time Frame: 24 hours
Population: This initial phase of the study was a pilot assessment of participants with bone sarcomas compared to participants with osteomyelitis.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Bone Sarcomas: Participants with bone sarcomas (osteosarcomas and Ewing sarcomas) evaluated with ferumoxytol-enhanced MRI.
- Osteomyelitis: Participants with osteomyelitis evaluated with MRI with ferumoxytol enhancement.
Arm/Group | Bone Sarcomas | Osteomyelitis
Number analyzed (Participants) | 5 | 4
milliseconds | 7.3 (1.9) | 7.7 (1.9)

2. Secondary Outcome: Differentiation of Bone Sarcomas Pre-ferumoxytol and Post-ferumoxytol Contrast
Description: Differentiation of bone sarcomas pre-ferumoxytol and post-ferumoxytol contrast was assessed by difference of mean T2 * relaxation time pre-ferumoxytol and post-ferumoxytol contrast, in bone sarcoma subjects only.
Time Frame: Baseline and Post-Treatment-24 hours
Population: Only the participants with bone sarcomas were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Bone Sarcomas Pre-ferumoxytol & Post-ferumoxytol Contrast: Participants with bone sarcomas (osteosarcomas and Ewing sarcomas) only.
Arm/Group | Bone Sarcomas Pre-ferumoxytol & Post-ferumoxytol Contrast
Number analyzed (Participants) | 10
milliseconds
  Pre-treatment: number analyzed (Participants) | 5
  Pre-treatment | 13.80 (2.80)
  Post-treatment | 8.27 (2.12)

3. Secondary Outcome: Differentiation of Lymphoma and Bone Sarcomas With Ferumoxytol-enhanced MRI
Description: Differentiation of lymphoma from bone sarcoma was assessed as the difference of mean T2 * relaxation time determined by ferumoxytol-enhanced MRI.
  .
Time Frame: 24 hours
Population: The analysis population for this outcome includes the participants with bone sarcoma who participated in the pilot study.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Mean T2 * Relaxation Time for Lymphoma Participants: Participants with lymphoma evaluated with ferumoxytol-enhanced MRI
- Mean T2 * Relaxation Time for Bone Sarcoma Participants: Participants with bone sarcoma, evaluated with ferumoxytol-enhanced MRI
Arm/Group | Mean T2 * Relaxation Time for Lymphoma Participants | Mean T2 * Relaxation Time for Bone Sarcoma Participants
Number analyzed (Participants) | 7 | 10
milliseconds | 14.83 (1.03) | 7.71 (0.60)

4. Secondary Outcome: Differentiation of CD68-positive Tumor-associated Macrophages (TAM) in Lymphomas and Bone Sarcomas
Description: Differentiation of CD68-positive tumor-associated macrophages (TAM) between lymphoma and bone sarcoma was assessed as the difference of mean area density of CD68-positive TAM in those populations.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Percentage of CD68-positive TAM
Groups:
- Mean Area Density of CD-68-positive TAM in Lymphoma: CD-68-positive tumor-associated macrophages (TAM) assessed in Lymphoma participants
- Mean Area Density of CD-68-positive TAM in Bone Sarcomas: CD-68-positive Tumor associated macrophages(TAMs)in Bone Sarcomas participants
Arm/Group | Mean Area Density of CD-68-positive TAM in Lymphoma | Mean Area Density of CD-68-positive TAM in Bone Sarcomas
Number analyzed (Participants) | 7 | 10
Percentage of CD68-positive TAM | 4.8 (1.2) | 6.1 (2.3)

5. Secondary Outcome: Differentiation of CD163-positive Tumor-associated Macrophages (TAM) in Lymphomas and Bone Sarcomas
Description: Differentiation of CD163-positive tumor-associated macrophages (TAM) between lymphoma and bone sarcoma was assessed as the difference of mean area density of CD163-positive TAM in those populations.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Percentage area of CD163-positive TAM
Groups:
- Mean Area Density of CD163-positive TAM in Lymphoma: CD163-positive tumor-associated macrophages (TAM) was assessed in participants with lymphoma
- Mean Area Density of CD163-positive TAM in Bone Sarcoma: CD163-positive tumor-associated macrophages (TAM) was assessed in participants with bone sarcomas
Arm/Group | Mean Area Density of CD163-positive TAM in Lymphoma | Mean Area Density of CD163-positive TAM in Bone Sarcoma
Number analyzed (Participants) | 7 | 10
Percentage area of CD163-positive TAM | 1.9 (1.5) | 9.4 (3.1)

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Feraheme: Intravenous injection of Feraheme, 5 mg Fe/kg
  Feraheme: 5 mg Fe/kg iv
  MR Scan: Standard of Care
Arm/Group | Feraheme
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feraheme (N=21)
Allergic reaction (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-04-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT01336803/Prot_SAP_000.pdf